CLINICAL TRIAL: NCT06972394
Title: Should Videolaryngoscopy Enter Routine Use? Unanticipated Difficult Airway: A Five-Year Experience in a Tertiary Care Hospital
Brief Title: Videolaryngoscopy at Unanticipated Difficult Airway
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-124
Record Dates: First submitted 2025-05-02; First posted 2025-05-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Difficult Airway; Videolaryngoscopy
Keywords: Anesthesia; intubation; airway management; laryngoscopy; difficult airway; videolaryngoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unanticipated difficult airway: In the present study, the records of patients with unanticipated difficult airway in the clinic were retrospectively reviewed. The aim was to compare the effects of direct laryngoscopy and videolaryngoscopy on glottic visualization, intubation success, and complications in patients with unanticipated difficult airway.

SUMMARY:
Glottic visualization, intubation success, complications and accidental esophageal intubation rate of direct laryngoscopy (DL) and videolaryngoscopy (VL) were compared in patients with UDA.

DETAILED DESCRIPTION:
Ethical approval for this study was obtained from the Clinical Research Ethics Committee of Tokat Gaziosmanpaşa University (25-MOBAEK-124). Data were collected by reviewing hospital automation systems, patient records, and difficult airway forms for patients who underwent elective surgery under general anesthesia and experienced unanticipated difficult airway (UDA) between January 2020 and March 2025. Patients with incomplete data, a prior history of difficult airway, or preoperative findings indicating a difficult airway were excluded from the study. Demographic variables-including age, gender, body mass index, comorbidities, and ASA scores-as well as airway examination findings such as Mallampati scores and Cormack-Lehane grades, were analyzed. Additionally, intubation methods, instruments used, and challenges encountered during airway management were evaluated. The effects of direct laryngoscopy (DL) and videolaryngoscopy (VL) on glottic visualization, intubation success, and complication rates were also compared.

In the relevant clinic, preoperative airway evaluation is performed by assessing the Mallampati classification, thyromental distance, sternomental distance, inter-incisor gap and angle, neck circumference, atlanto-occipital joint mobility, upper lip bite test, retrognathia, prominent upper incisors, high and narrow palate, macroglossia, hoarseness, dyspnea on exertion, and history of difficult airway. In patients without any predictors of difficult airway, routine intubation is performed using DL in the sniffing position. The management of patients with UDA is conducted according to a specific institutional protocol. In appropriate cases where mask ventilation and oxygenation can be maintained, a hyper-angulated C-MAC® D-Blade videolaryngoscope (Karl Storz, Tuttlingen, Germany) is used as a rescue technique in patients who cannot be intubated using DL. If tracheal intubation cannot be achieved with videolaryngoscopy or other methods and the patient is awakened, and if the surgical procedure still requires general anesthesia, awake intubation using fiberoptic bronchoscopy (FOB) is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years
* Patients with unanticipated difficult airway

Exclusion Criteria:

* Patients with missing data
* Patients with a history of difficult airway
* Patients with signs of difficult airway on preoperative evaluation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients with no signs of difficult airway (unanticipated difficult airway) in preoperative evaluation will be investigated retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Intubation success | From anesthesia induction until the attempt of intubation is completed (peri-induction period).
  Successful intubation rate with DL or VL in patients with unpredictable difficult airway

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Preoperative airway findings of patients, devices used in airway management and their results and complications
Supporting Information: Study Protocol, SAP
Time Frame: January 2020 and March 2025
Access Criteria: The data used to support the findings of this study can be obtained from the corresponding author on request.